CLINICAL TRIAL: NCT03816618
Title: The Healing Effects Of Honey and Hydrogel Products On The Diabetic Foot
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cyberjaya University College of Medical Sciences (Other)
Collaborators: Diabetic Center-KFSH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CyberjayaU
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Foot
Keywords: purilon gel; medihoney; fucidine
MeSH Terms: conditions — Diabetic Foot | interventions — Hydrogels

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CONTROL (Experimental): CONTROL GROUP
  Interventions: Drug: Fucidin Ointment
- TREATMENT1 (Experimental): TREATMENT GROUP 1
  Interventions: Drug: Medihoney Gel in A Tube
- TREATMENT2 (Experimental): TREATMENT GROUP 2
  Interventions: Drug: Hydrogel
- TREATMENT3 (Experimental): TREATMENT GROUP 3
  Interventions: Drug: Medihoney Gel in A Tube; Drug: Hydrogel

INTERVENTIONS:
Drug: Medihoney Gel in A Tube — TREATMENT1
  Other Names: MEDIHONEY
  Arms: TREATMENT1; TREATMENT3
Drug: Hydrogel — PURLOIN GEL
  Other Names: PURLOIN
  Arms: TREATMENT2; TREATMENT3
Drug: Fucidin Ointment — FUCIDIN ANTIBIOTIC OINTMENT 10%
  Other Names: FUCIDIN OINTMENT 10%
  Arms: CONTROL

SUMMARY:
The Healing effects of Honey and Hydrogel Products on the Diabetic Foot.

Abstract:

Diabetes mellitus epidemiology is increasing dramatically affecting high numbers of the world's population, one of the highest risk consequences is diabetic foot and which might lead to leg amputation causing a permanent disability for the patient.

Several studies had been conducted on the options available to treat diabetic foot ulcer, Honey products and Hydrogel stands out as an effective topical treatment for the foot ulceration.

This study discusses the effectivity rate of these products and compares it with the classical methods followed to treat DF using topical and systematic antibiotics.

Hence; our research raises the following questions:

1. What is the effect of Honey and Hydrogel on the foot anatomy and physiology of DF patients?
2. Could the investigators introduce a new protocol to treat DF using Honey and Hydrogel products?

Aiming to achieve the following objects:

1. To provide a new protocol to improve the anatomy and physiology of DF.
2. To compare the efficacy of combined Hydrogel and Honey products on the diabetic foot ulcer.

Reaching there the investigators are expecting to:

1. To compare the healing time between the patients treated with hydrogel/honey products and the control treatment patients.
2. To compare Lab parameters improvements between the patients treated with hydrogel/honey products and the control treatment patients.
3. To compare neurological improvements between the patients treated with hydrogel/honey products and the control treatment patients.
4. To compare the anatomical improvements between the patients treated with hydrogel/honey products and the control treatment patients.

In order to provide a clear estimation for the safety and effectivity profile for each treatment method.

Based on that the investigators are conducting using single blinded randomized clinical trial

Suggesting the following Hypothesis: Treatment using topical MediHoney gel and/or Hydrogel together separately in association with empiric antibiotic regimens have a higher success rate comparing with treatment using topical and empiric antibiotic.

A total of 120 DM patients from Outpatients DM type 2 will be included in this study, following up at diabetic foot center Al-Qaseem Saudi Arabia. Patients will be divided into 4 groups:

1. st group will be treated with topical Medihoney product and empiric antibiotic.
2. nd group will be treated with topical Hydrogel (purloin) gel and empiric antibiotic.
3. rd group will be treated with a combination of Medihoney gel and Hydrogel (purloin) gel and empiric antibiotic.

The 4th group will be treated with a combination of systematic and topical fucidin 1% antibiotic this group will be a controlled group.

Based on the expected results the investigators are estimating that this study will raise the awareness of both health care personnel and the diabetic patients about this condition. It is expected to provide a clear efficacy estimation for each treatment method followed, facilitating the choice of treatment for physicians.

DETAILED DESCRIPTION:
The Healing Effects of Honey and Hydrogel Products on the Diabetic Foot. Title 1 TITLE OF RESEARCH PROPOSAL: THE HEALING EFFECTS OF HONEY AND HYDROGEL PRODUCTS ON THE DIABETIC FOOT.

Trial registration 2a Registration by clinical trial. gov, by PRS password available and got approval Number H-04-Q-001 from National Committee of Bio & Med. Ethics(NCBE).

Protocol version 3 Protocol version helps to mitigate potential confusion over which will be started after the ethical approval.

Funding 4 The treatment packs will be prepared by diabetic foot centre, materials: natural drugs, (medihoney gel and purloin gel and fucidine ointment 1%) placebo.

Roles and responsibilities 5a Prof. Dr. Husni Al-Goshae [PHD Neuroscience (UK)], Prof. Dr. Hamdan Noor [PHD Ox Ford University Physiologist], Consultant Dr. Hamad Saleh Alshubrumi [Endocrinologist King Fahad Specialist Hospital, Al-Qassim, KSA].

5b Trial Sponsor: Cyberjaya University College of Medical Science Address: Persiaran Bestari Cyber11, 63000, Cyberjaya, Selangor Malaysia Telephone: 0060383137000 Website: www.cybermed.edu.mi

5c This funding source had no role in the design of this study and will not have any role during its execution, analyses, interpretation of the data, or decision to submit results.

5d Design and conduct for preparation of protocol and revisions, investigators brochure and publication of study reports.

Trial management committee (TMC) Principle [sic] investigator, research physician, administrator) Study planning , Organization of steering committee meetings Provide annual risk report MHRA [Medicines and Healthcare Products Regulatory Agency] and ethics committee, SUSAR [Serious unexpected suspected adverse events] reporting to MHRA and Roche Responsible for trial master file, Budget administration and contractual issues with individual centers , Advice for lead investigators Audit of 6 monthly feedback forms and decide when site visit to occur.

Assistance with international review, board/independent ethics committee applications; Data verification Randomization

Introduction Background and rationale 6a Outpatient DM type 2 patients follow up at diabetic foot center adult more or equal 18 years).

Research question :

1. - What is the effect honey and hydrogel on the foot anatomy and physiology of DF patients?
2. - Could the investigators introduce a new protocol to treat DF? the investigators find it very necessary to define the real rate for these two agents treating DF ulcers , to establish clear clinical evidence supporting the prefer ability of using such natural low risk and relatively low cost agents in the treatment plan comparing with the use of the classical antibiotic treatment .

6b "Choice of comparator Effectivity of each product treating DF, the investigators find it more beneficially to establish a comparative study between such safe and low cost products and antibiotics recommending a less complicated and safe treatment method using honey and /or hydrogel rather than depending on the classic antibiotic method with all of its potential contraindications and restrictions in sensitive group of patients such as DM patients".

Objectives 7 Research hypothesis Treatment using topical MediHoney gel and/or Hydrogel together or separately in association with empiric antibiotic regimens have a higher success rate comparing with treatment using topical and empiric antibiotic.

Study Objectives Main Objectives a) To provide a new protocol to improve to anatomical and physiological response of DF.

b) To compare the efficacy of combined hydrogel and honey products on DF ulcer.

Specific objectives:

1. To compare the healing time between the patients treated with hydrogel/honey products and the control treatment patients.
2. To compare Lab parameters improvements between the patients treated with hydrogel/honey products and the control treatment patient such as CSR and WBC, etc.
3. To compare neurological improvements between the patients treated with hydrogel/honey products and the control treatment patients.
4. To compare the anatomical improvements between the patients treated with hydrogel/honey products and the control treatment patients.

   8 The study will be conducted using single blinded randomized clinical trial from October 2018 to February 2021, it will be conducted on DF patients with any stage of diabetic foot ulcer in the Center of Diabetic Foot, King Fahad specialist hospital Al-Qassim KSA.

   Randomization will be performed as block randomization with a 1:3 allocation.

   Methods: Participants, interventions, and outcomes Study setting 9 Outpatients DM type 2 patients, follow up at diabetic foot center. Centre of diabetic foot, King Fahad Specialist Hospital Al- Qassim KSA.

   Eligibility criteria 10 1.1.1. Inclusion Criteria:

   It is mandatory for all of the participants to follow each of the following criteria:
   * Adult more or equal 18 years with type 2 DM.
   * Diagnosed with stable DF with any stage of foot ulcer

   Exclusion Criteria:

   • Patients with unstable severe conditions who requires hospitalization.

   • Patients with incomplete data and those who decided to withdraw.
   * Read and understood the consent of the research and didn't approve to participate accordingly.
   * Patients with open osteomyelitis with discharged us.
   * DM patients with ischemic peripheral PAD gangrene.
   * Charcoat diabetic foot CDF.

   Interventions 11a Patients will be divided into 4 groups:

   1st group will be treated with topical Medihoney gel product and empiric antibiotic (systematic) until the result of culture swab wound appears.

   2nd group will be treated with topical Hydrogel (purloin) gel and empiric antibiotic (systematic) until the result of culture swab wound appears.

   3rd group will be treated with a combination of topical Medihoney gel and Hydrogel (purloin) gel and empiric antibiotic (systematic) until the result of culture swab wound appears.

   The 4th group will be treated with a combination of systematic and topical Fucidin ointment 1% and empiric antibiotics, (systematic) this group will be a controlled group until the result of culture swab wound appears.

   11b Medihoney Gel, Purloin Gel, Fucidin Ointment 1% placebo drug 11c All groups will be monitored and the prospects for clinical, neurological, and anatomical, improvements will be followed up by the laboratory.

   11d For 3-12 weeks: Close observation and monitoring the topical treatment

   Appearance of ischemic arterial disease during participation Contraindication Treatment DFU(Allergic) As well as termination of participant

   Outcomes 12 Main Outcome Measurement:

   Ulcer size • Baseline: Size of the Ulcer before the beginning of treatment • Size will be monitored upon the commencement of the treatment until reaching the healing condition.

   • Main measurement: Time needed to reach the condition of fully healing of the ulcer (ULCER SIZE IS ZERO) Participant timeline 13 Dressing patient daily. Measurement of wound every week. This will continue for 3-12 weeks with DF patients. Sample size 14 Sample size calculation

   Studies that are analyzed by chi-square or Fisher's exact test calculated sample size with professor statistical in the CUCMS

   Alpha is 5% Estimated power of the study: 80% Ratio of unexposed to exposed 3 (3 groups of treatment to 1 control group) Expected of unexposed with outcome incidence Expected exposed with outcome incidence

   The sample size formula without the correction factor by Fleiss is:

α: The probability of type I error 5% β: The probability of type II error 20% Zalpha/2=1.96 Zbetta/2=0.842 P0: The proportion of people with control treatment applied in population 1 (0.70) P1: The proportion of people with random treatment applied in population 3 (0.95) r: The ratio of unexposed to exposed 0.33 NFleiss: Required sample size for the population 1 using Fleiss formula According to the equation N Fleiss should be 30 per group patients.

Recruitment 15 Targeted Sample size:

Our sample size will be 120 patients (due to possibility and cost effectivity) designed as 30 patients in each group.

Methods: Assignment of interventions (for controlled trials)

Allocation: Matching will be done depending on 3 variables:

* Gender:
* Age:
* Dounis classification:

Type I Type II Type III (A,B,C)

Sequence generation 16a Participants will be randomly assigned to either control or experimental group with a 1:3 allocation

Type of randomization: single, blind randomization convenient for all patients follow up in the DF center, with matching factors; age, gender, Dounis anatomical classification.

Allocation concealment mechanism 16b Participants will randomised using central randomisation service. Allocation concealment will be ensured, as the service will not release the randomization code until the patient has been recruited into the trial, which takes place after all baseline measurements have been completed.

Implementation 16c All patients who give consent for participation and who fulfil the inclusion criteria will be randomized. Randomization will be requested by the staff member responsible for recruitment and clinical interviews from CenTrial [Coordination Centre of Clinical Trials]. In return, CenTrial will send an answer form to the study therapist who is not involved in assessing outcome of the study. This form will include a randomization number. In every center closed envelopes with printed randomization numbers on it are available. For every randomization number the corresponding code for the therapy group of the randomization list will be found inside the envelopes. The therapist will open the envelope and will find the treatment condition to be conducted in this patient. The therapist the gives the information about treatment allocation to the patient. Staff responsible for recruitment and symptom ratings is not allowed to receive information about the group allocation.

Blinding (masking) 17a Due to the nature of the intervention, participants can be blinded to allocation but are strongly inculcated not to disclose the allocation status of the participant at the follow up assessments. An employee outside the research team will feed data into the computer in separate datasheets so that the researchers can analyze data without having access to information about the allocation.

17b If un-blinding is deemed to be necessary, the investigator should use the system for emergency un-blinding through the local emergency number as the back-up system.

Methods: Data collection, management, and analysis Data collection methods 18a Plans for assessment and collection of outcome, baseline, and other trial data, including any related processes to promote data quality (eg, duplicate measurements, training of assessors) and a description of study instruments (eg, questionnaires, laboratory tests) along with their reliability and validity, if known. Reference to where data collection forms can be found, if not in the protocol

Main Outcome Measurement:

Ulcer size • Baseline: Size of the Ulcer at the before the beginning of treatment

• Size will be monitored upon the commencement of the treatment until reaching the healing condition.

• Main measurement: Time needed to reach the condition of fully heal of the ulcer (ULCER SIZE IS ZERO) Quality Control of the Core Lab Data from the Core Lab will be securely transmitted in batches and quality controlled in the same manner as Core Coordinating Center Data.

18b Provide written feedback to all patients about the results of the health screening. Maintain interest in the study through materials and mailing. Send letters to patients prior to the final data collection, reminding them of the upcoming data collection.

Participants may withdraw from the study for any reason at any time. The investigator also may withdraw participants from the study in order to protect their safety and/or if they are unwilling or unable to comply with required study procedures after consultation with the protocol chair.

Data management 19 Participant files are to be stored in numerical order and stored in a secure and accessible place and manner. Participant files will be maintained in storage for a period of 3 years after completion of the study.

Weekly reports with information on missing data, missing forms, and missing visits. Personnel at the Core Coordinating Center and the Participating Sites should review these reports for accuracy and report any discrepancies to the investigator.

Statistical methods 20a Statistical methods for analyzing primary and secondary outcomes. Reference to where other details of the statistical analysis plan can be found, if not in the protocol

Analysis methods will depend on the improvements according to Dounis classification, as well as each of the clinical, neurological, anatomical, and angiographic improvement rate.

20b Methods for any additional analyses (eg, subgroup and adjusted analyses)

The data will be analyzed using version 23 of SPSS statistical software (SPSS Inc., Chicago, IL, USA). Descriptive statistics will be calculated as proportions or as means (with standard deviations) as appropriate. The significance level will be set as p value<0.05.

20c The investigators propose declaring medical management non-inferior to interventional therapy, only if shown to be non-inferior using both the "intention to treat" and "per protocol" analysis sets.

Methods: Monitoring Data monitoring 21a The DMC is independent of the study organizers. During the period of recruitment to the study, interim analyses will be supplied, in strict confidence, to the DMC, together with any other analyses that the committee may request. This may include analyses of data from other comparable trials.

21b An interim-analysis is performed on the primary endpoint when 50% of patients have been randomized and have completed the 6 months follow-up.

Harms 22 Adverse events will be collected after the subject has provided consent and enrolled in the study. If a subject experiences an adverse event after the informed consent document is signed (entry) but the subject has not started to receive study intervention.

Auditing 23 The quality and completeness of the data will be reflective of the state of the art in clinical trials. The focus of the visit/electronic monitoring will be on source document review and confirmation of adverse events. The monitor will verify the following variables for all patients: initials, date of birth, sex, signed informed consent, eligibility criteria, date of randomization, treatment assignment, adverse events, and endpoints.

Ethics and dissemination Research ethics approval 24 The protocol, site-specific informed consent forms (local language and English versions), participant education and recruitment materials, and other requested documents-and any subsequent modifications - also will be reviewed and approved by the ethical review bodies.

The Investigator will make safety and progress reports and summaries review of safety and/or efficacy.

Protocol amendments 25 Any modifications to the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, patient population, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol.

Consent or assent 26a Trained Research Nurses will introduce the trial to patients who will receive information sheets. Research Nurses will discuss the trial with patients in light of the information provided in the information sheets. Patients will then be able to have an informed discussion with the participating consultant. Research Nurses will obtain written consent from patients willing to participate in the trial. Information sheets and consent forms are provided for all parents involved in the trial

26b A materials consent will be obtained to specifically address the collection

Confidentiality 27 All study-related information will be stored securely at the study site. All participant information will be stored in locked file cabinets in areas with limited access. All laboratory specimens, reports, data collection, process, and administrative forms will be identified by a coded ID [identification] number only to maintain participant confidentiality. All records that contain names or other personal identifiers, such as locator forms and informed consent forms, will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems. Forms, lists, logbooks, appointment books, and any other listings that link participant ID numbers to other identifying information will be stored in a separate, locked file in an area with limited access.

Declaration of interests 28 He does not have any paid consultancies with pharmaceutical companies, and is not a member of the Speaker's Panel of any company.

Access to data 29 All Principal Investigators will be given access to the cleaned data sets. Project data sets will be housed on the Project Accept Web site and/or the file transfer protocol site created for the study, and all data sets will be password protected. Project Principal Investigators will have direct access to their own site's data sets, and will have access to other sites data by request. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information

Ancillary and post-trial care 30 The liability of the manufacturer is strictly limited to those claims arising from faulty manufacturing of the commercial product and not to any aspects of the conduct of the study.

Dissemination policy 31a The Publications subcommittee will review all publications following the guidelines and report its recommendations to the Steering Committee.

the scientific integrity of the project requires that the data from all BEST Evaluation of Survival Trial sites be analyzed study-wide and reported Each paper must be submitted to the appropriate Subcommittee for review of its appropriateness and scientific merit prior to submission.

31b There are three classes of reports;

a) Reports of the major outcomes of the study. b) Reports addressing in detail one aspect. c) Reports of data derived from a subset of centers.

31c Data sharing statement No later than 3 years after the collection of the 2-year post randomization interviews, The investigators will deliver a completely de-identified data set to an appropriate data archive for sharing purposes Appendices Informed consent materials 32 Study number: Not available Investigator Name: Dr. Wael Searan Address: Center Endocrinology and Diabetes, Buraidah, Al-Qassim, KSA. Consent Form: This consent form is part of the informed consent process. It is designed to give you an idea of what this research study is about and what will happen to you if you choose to be in the study…

Biological specimens 30

In my study measurement there is no any biological specimens.

ELIGIBILITY:
Inclusion Criteria:

* Adult more or equal 18 years with type 2 DM.
* Diagnosed with stable DF with any stage of foot ulcer

Exclusion Criteria:

* Patients with unstable severe conditions who requires hospitalization.
* Patients with incomplete data and those who decided to withdraw.
* Read and understood the consent of the research and didn't approve to participate accordingly.
* Patients with open osteomyelitis with discharged us.
* DM patients with ischemic peripheral PAD gangrene.
* Charcoat diabetic foot CDF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Ulcer size | FROM 3 WEEKS UP TO 12 WEEKS
  ULCER SIZE

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Diabetic Center-KFSH, Buraidah, Al-Qassim
  - Diabetes Center, Center Diabetic Foot, King Fahd Specialist Hospital, Ministry Of Health Buraydah; Al Qassim; Saudi Arabia, Buraidah, Elqassim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — https://www.nice.org.uk/guidance/CG10 — National Institute for Health and Clinical Excellence. Type 2 diabetes; prevention and management of foot problems